CLINICAL TRIAL: NCT00887640
Title: Impact of Temsirolimus Therapy on Circulating Tumor Cell Biology In Men With Castration Resistant Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016256
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: metastatic; Temsirolimus; prostate; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — temsirolimus; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temsirolimus 25 mg (Experimental): Temsirolimus 25mg was administered by IV infusion each week (days 1, 8, 15, and 22 of each 28 day cycle). The infusion was to be administered over a period not less than 30 minutes and was to be completed within 60 minutes. Subjects were premedicated with 25 to 50 mg IV or PO diphenhydramine (or an alternative antihistamine in case of allergies) 30 minutes prior to the infusion.
  Interventions: Drug: Temsirolimus; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Temsirolimus — dosage form: IV dosage, frequency and duration: 25mg weekly until clinical progression
  Other Names: Torisel
Drug: Diphenhydramine — Dosage form: IV or PO Dosage, frequency and duration: 25-50mg, 30 minutes prior to Temsirolimus infusion
  Other Names: Benadryl

SUMMARY:
This is a single arm study of 11 men with treatment refractory metastatic Castrate Resistant Prostate Cancer (CRPC) who will receive temsirolimus IV at a dose of 25 mg weekly until progression. Progression will not include Prostate Specific Antigen (PSA) progression; however, upon PSA progression, the addition of an anti-androgen will be permitted. The primary objective of the study is to evaluate change in circulating tumor cell (CTC) counts over time in men with metastatic treatment-refractory CRPC in response to temsirolimus therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoma of the prostate. Histologic evidence may be confirmed through local or metastatic biopsy review
* Radiographic Evidence of metastatic disease
* Evidence of disease progression despite castrate levels of testosterone.
* A circulating timor cell count using FDA approved CellSearch methodology of ≥ 10 per 7.5 cc whole blood, drawn within 4 weeks of study registration
* Serum PSA greater than or equal to 2ng/dl at registration
* At least 4 weeks since prior palliative radiation therapy and/or major surgery, and resolution of all toxic effects of prior therapy NCI Common Toxicity Criteria for Adverse Effects (CTCAE) Grade less than or equal to 1
* Age ≥ 18 years
* Adequate laboratory parameters
* Karnofsky Performance Status ≥ 60
* Life expectancy of at least 3 months

Exclusion Criteria:

* History of or active central nervous system metastases
* The use of cytotoxic, biologic, or hormonal therapies within 4 weeks of study entry.
* Subjects receiving known strong Cytochrome P450 3A4 (CYP3A4) isoenzyme inhibitors and/or inducers
* Major surgery, open biopsy, traumatic injury, or radiotherapy within 4 weeks of the screening visit
* Have not recovered from prior biopsy, surgery, traumatic injury, and/or radiation therapy.
* Presence of non-healing wound or ucer
* Grade ≥ 3 hemorrhage in the past month to study entry
* Hypertension with systolic blood pressure of ≥ 180 mmHg and/or diastolic pressure ≥ 100 mmHg (Anti-hypertensive medications are permitted)
* Subjects with Class 2-4 heart disease or any history of congestive heart failure with an ejection fraction <50% or a recent (within 12 months) cardiovascular event.
* Anticoagulation with warfarin
* Diabetes mellitus with glycosylated hemoglobin A1c ≥ 10% despite therapy
* History of interstitial pneumonitis
* Subjects with active autoimmune disorder(s) being treated with immunosuppressive agents within 4 weeks prior to screening visit
* Subjects receiving immunosuppressive agents and those with chronic viral/bacterial/fungal illnesses. Replacement doses of corticosteroids are permitted.
* Active infection(s), active antimicrobial therapy or serious intercurrent illness.
* History of other prior malignancy in past 5 years, other than basal cell carcinoma, squamous cell carcinoma of the skin, cervical carcinoma in sity, localized prostate cancer, or superficial bladder cancer.
* Agreement to use medically acceptable contraceptive methods while on study and for 3 months after the last dose of temsirolimus.
* Any other major medical or psychiatric illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study, including inability to absorb oral medications.
* Known hypersensitivity to any of the components in the temsirolimus infusion or other medical reasons for not being able to receive adequate premedication.
* Corrected QT interval on baseline EKG of >500 milliseconds
* the use of agents that significantly prolong the Corrected QT interval and who are unable to stop medications prior to study initiation.
* Prior exposure to an Mammalian Target of Rapamycin (mTOR) inhibitor
* Presence of nephrotic syndrome as determined by clinical evaluation of 24 hour urine.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, ScM, Principal Investigator — Duke Unversity Medical Center
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Virginia Oncology Associates, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temsirolimus 25 mg
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 61 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Circulating Tumor Cell (CTC) Counts in Men With Metastatic Treatment-refractory Castration-resistant Prostate Cancer.
Description: Median percent change in CTC count from baseline to 8 weeks of treatment. Percent change was calculated by determining the percentage increase or decrease in CTC count from baseline.
Time Frame: Baseline to 8 weeks
Population: CTC count at both baseline and week 8 were assessable in 8 of the 11 patients as CTCs were collected at both time points in these patients. Missing CTC data for 3 of the 11 patients due to laboratory error or no CTC available at various time points.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 8
percent change | -20 [-53 to 73]

2. Secondary Outcome: Percent Change in CTC Count From Baseline to 12 Weeks of Treatment.
Description: To evaluate the change in CTC counts upon the addition of an anti-androgen upon PSA progression while on temsirolimus therapy
Time Frame: Baseline to 12 weeks
Population: Data were insufficient to evaluate this outcome. Outcome not available at 12 weeks. CTCs were not collected at week 12 and thus were not analyzed.
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Mean Percent of N-cadherin Expression at Baseline and 8 Weeks of Treatment.
Description: Measures of epithelial plasticity on CTCs in response to Mammalian Target of Rapamycin (mTOR) inhibition with temsirolimus, using genomic and protein immunohistochemical methodology. N-cadherin was measured in CTCs captured using the CellSearch profile kit. The proportion of CTCs expressing N-cadherin was calculated and divided by the total number of CD45-negative, pan cytokeratin (CK) - positive, and 4',6-diamidino-2-phenylindole (DAPI+) intact cells to give a fractional expression of N-cadherin. Results are reported as a percentage.
Time Frame: Baseline and 8 weeks
Population: N-cadherin expression at both baseline and 8 weeks was evaluable in 7 patients.
Measure: Median (Full Range); unit: Percent expression
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 7
Percent expression
  Expression at baseline | 91 [65 to 100]
  Expression at 8 weeks | 92 [50 to 100]

4. Secondary Outcome: Percent Change in LDH
Description: To evaluate and correlate changes in serum Lactate Dehydrogenase (LDH) with CTC count changes over time in men with Castrate Resistant Prostate Cancer (CRPC) treated with temsirolimus
Time Frame: Baseline to 12 weeks
Population: Data were insufficient to evaluate this outcome. Data not collected. This outcome was not performed due to availability and feasibility of the tests involved.
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to Prostate Cancer Clinical Trial Working Group 2 (PCWG2) criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Additionally, according to PCWG2 criteria, disease progression in bone is defined as 2 or more new lesions seen on bone scan compared with the baseline scan used for trial entry. Per PCWG2 guidelines, therapy was not discontinued solely due to a rise in PSA alone.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 11
Months | 1.9 [0.9 to 3.1]

6. Secondary Outcome: Maximum Rate of Change of Prostate-Specific Antigen (PSA).
Description: Percent change in PSA between baseline and the measurement time point where the largest change in PSA occurred. Note that a positive change (greater than 0) indicates an increase in PSA, and a negative change (less than 0) indicates a decrease.
Time Frame: Baseline to 7 months
Measure: Median (Full Range); unit: Percent change
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 11
Percent change | 48 [-32 to 954]

7. Secondary Outcome: Time to PSA Progression
Description: Time in months from the start of study treatment to the date of first PSA progression . Patients alive who had not progressed as of the last follow-up or patients who had expired had time to PSA progression censored at the last follow-up date or death date. The median was estimated using a Kaplan-Meier curve.
Time Frame: 2 years
Population: Data were insufficient to evaluate this outcome. Data not collected. PSA responses were not observed in this study and PSA progression dates would essentially be the same as the radiographic PFS dates.
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Time to Second PSA Progression After Addition of Anti-androgen Therapy
Description: Time in months from the time of anti-androgen therapy to the date of second PSA progression . Patients alive who had not progressed as of the last follow-up or patients who had expired had time to second PSA progression censored at the last follow-up date or death date. The median was estimated using a Kaplan-Meier curve.
Time Frame: 2 years
Population: Data were insufficient to evaluate this outcome. Data not collected. Patients progressed radiographically before 2nd PSA progression occurred.
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 0

9. Secondary Outcome: Change Over Time in CTC Gene Expression Profile
Description: Percent change in CTC gene expression from baseline to 8 or 12 weeks of treatment.
Time Frame: 12 weeks
Population: as for outcome 4
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Safety and Tolerability of Temsirolimus
Description: Total number of grade 3, 4, and 5 adverse events at least possibly related to temsirolimus therapy. Adverse events were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 and were converted to 4.0 for the purposes of reporting to ClinicalTrials.gov.
Time Frame: 2 years
Measure: Number; unit: Adverse Events
Arm/Group | Temsirolimus 25 mg
Number analyzed (Participants) | 11
Adverse Events
  Grade 3 Adverse Events | 28
  Grade 4 Adverse Events | 2
  Grade 5 Adverse Events | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov
Arm/Group | Temsirolimus 25 mg
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus 25 mg (N=11)
Anemia (Blood and lymphatic system disorders) | 1
Lung infection- Pneumonia (Infections and infestations) | 1
Stroke- Hemorrhagic (Nervous system disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Vascular disorders - Subdural Hemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus 25 mg (N=11)
Anemia (Blood and lymphatic system disorders) | 5
Palpitations (Cardiac disorders) | 1
Night blindness (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Lip Swelling (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 6
Fever (General disorders) | 3
Pain (General disorders) | 1
Eye Infection (Infections and infestations) | 1
Infection - Picc Line (Infections and infestations) | 1
Lung infection- Pneumonia (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Alkaline phosphatase increased (Investigations) | 1
Creatinine increased (Investigations) | 3
INR increased (Investigations) | 1
Investigations - Fluid Overload (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Weight Loss (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypoalbuminenima (Metabolism and nutrition disorders) | 1
Hypocalcinemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponaturemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Pain - Lower Extremities Bilateral (Musculoskeletal and connective tissue disorders) | 1
Pain, Intermittant- Lower Left Quadrant (Musculoskeletal and connective tissue disorders) | 1
Pain- Bilateral Jaw (Musculoskeletal and connective tissue disorders) | 1
Pain- Bone (Musculoskeletal and connective tissue disorders) | 1
Pain- Left Femur (Musculoskeletal and connective tissue disorders) | 1
Pain- Left Hip / Low Back (Musculoskeletal and connective tissue disorders) | 1
Pain- Left Hip / Thigh (Musculoskeletal and connective tissue disorders) | 1
Pain- Left Shoulder (Musculoskeletal and connective tissue disorders) | 1
Pain- Left Side (Musculoskeletal and connective tissue disorders) | 1
Pain- Right Flank (Musculoskeletal and connective tissue disorders) | 1
Pain- Right jaw (Musculoskeletal and connective tissue disorders) | 1
Pain- left flank area (Musculoskeletal and connective tissue disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 1
Nervous system disorders - Nightmares (Nervous system disorders) | 1
Nervous system disorders- Restless Legs (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Right hydonephrosis (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash - Groin (Skin and subcutaneous tissue disorders) | 1
Rash - Right Arm and Leg (Skin and subcutaneous tissue disorders) | 1
Rash- Ankles (Skin and subcutaneous tissue disorders) | 1
Rash- Penis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event- Pulmonary Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes